CLINICAL TRIAL: NCT03742947
Title: Study of Peripartum Haemostasis and Effects of Tranexamic Acid in Caesarean Delivery: Biologic Ancillary Study in TRAAP2 Patients Recruited at the Bordeaux University Hospital: BIO-TRAAP
Brief Title: Haemostasis and Tranexamic Acid in Caesarean Delivery
Acronym: BIO-TRAAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bordeaux Association for Training and Research in Obstetric Gynecology (Unknown); Association of Anesthesiologists and Intensivists of Vascular Surgery and Transplantation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CHUBX 2018/24
Record Dates: First submitted 2018-10-30; First posted 2018-11-15 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Postpartum Hemorrhage; Hyperfibrinolysis
Keywords: ancillary biologic study; fibrinolysis; tranexamic acid; post-partum haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Three blood samples of 20 ml each at T0 after the anesthesia for the caesarean section and before the administration of the product (TXA or placebo), T15 fifteen minutes after the administration of the product and T120, 2 hours after the administration of TRAAP2 study IMP (tranexamic acid or placebo).
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): intravenous administration of 10-mL of tranexamic acid (EXACYL® 1 g/10 ml I.V., solution injectable)
  Interventions: Diagnostic Test: peripartum haemostasis
- Chloride solution (Placebo Comparator): sodium intravenous administration of 10-mL of chloride solution (0.9% -10mL)
  Interventions: Diagnostic Test: peripartum haemostasis

INTERVENTIONS:
Diagnostic Test: peripartum haemostasis — Three blood samples of 20 ml each at T0 after the anaesthesia for the caesarean section and before the administration of the product (TXA or placebo), T15 fifteen minutes after the administration of the product and T120, 2 hours after the administration of the product.

SUMMARY:
The aim of the study is to evaluate haemostasis and fibrinolysis in peripartum of caesarean delivery and the effect of tranexamic acid (TXA) given in prevention of post-partum haemorrhage (PPH).

DETAILED DESCRIPTION:
Post-partum haemorrhage (PPH) remains a leading cause of maternal morbidity and mortality. Haemostasis and fibrinolysis are activated in peripartum. Fibrinolysis is decreased during pregnancy, is quickly activated after childbirth and can be overactivated in case of PPH. Tranexamic acid (TXA), an antifibrinolytic drug, has been proven to efficiently decrease bleeding and death in PPH. Its place in prevention of PPH after caesarean section remains to be established. The aim of the study protocol TRAAP2 is to conduct a large multicentre randomized, double blind placebo-controlled trial to adequately assess the impact of TXA for preventing PPH following a caesarean section. Peripartum is also a period of increased thrombo-embolic risk. TXA has never been proven to increase thromboembolic events. Nevertheless, it seems important to reserve TXA for women with activated fibrinolysis.

The aim of the ancillary biologic study BIO-TRAAP is thus to explore haemostasis and fibrinolysis in peripartum, to determine which women will in the future benefit from TXA. Fibrinolysis will be studied by clot lysis time by Global Fibrinolytic Capacity test on the Lysis Timer (GFC/LT), t-PA, PAI-1, PAI-2, euglobulin clot lysis time, plasminogen, plasmin-anti-plasmin complex, thrombin-anti-thrombin complex, fibrin degradation products (FDP).

ELIGIBILITY:
Inclusion Criteria:

* patient randomized into TRAAP2 study (NCT03431805):

  * adult women admitted for a planned caesarean delivery,
  * at term ≥ 34 weeks,
  * haemoglobin level at the last blood sample >9g/dl,
  * blood Formula numbering within 7 days before caesarean delivery, informed signed consent)
* informed signed consent for BIO-TRAAP

Exclusion Criteria:

* patient not included into TRAAP2 study:

  * previous thrombotic event or pre-existing pro-thrombotic disease,
  * epileptic state or history of seizures,
  * presence of any chronic or active cardiovascular disease outside hypertension,
  * any chronic or active renal disease including renal, chronic or acute insufficiency (glomerular flow <90mL / min), and chronic or active liver disease at risk thrombotic or haemorrhagic,
  * autoimmune disease,
  * sickle cell disease,
  * placenta praevia,
  * placenta accreta/increta/percreta,
  * abruption placentae,
  * eclampsia,
  * HELLP syndrome,
  * in utero fetal death,
  * administration of low-molecular-weight heparin or antiplatelet agents during the week before delivery,
  * general anaesthesia,
  * hypersensitivity to tranexamic acid or concentrated hydrochloric acid, instrumental extraction failure,
  * multiple pregnancy with genital delivery of the first twin and caesarean delivery for the second or at third trimester,
  * poor understanding of the French language

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Clot lysis time | Baseline (defined as the time of insertion of the peripheric venous line)
  Clot lysis time in minutes studied by the Global Fibrinolytic Capacity on the Lysis Timer

SECONDARY OUTCOMES:
Lysis Timer clot lysis time | Time 15min and Time 120min (defined as 15 minutes 120 minutes after the administration of the product, respectively)
  Clot lysis time in minutes studied by the Global Fibrinolytic Capacity on the Lysis Timer
Routine clot lysis time | Baseline, Time 15min, and Time 120min
  Clot lysis time in minutes studied by the routine biological tests
t-PA | Baseline, Time 15min, and Time 120min
  tissue-Plasminogen Activator (ng/ml)
PAI-1 | Baseline, Time 15min, and Time 120min
  Plasminogen activator inhibitor-1 (ng/ml)
PAI-2 | Baseline, Time 15min, and Time 120min
  Plasminogen activator inhibitor-2 (ng/ml)
Euglobulin clot lysis time | Baseline, Time 15min, and Time 120min
  Euglobulin clot lysis time (min),
Plasminogen | Baseline, Time 15min, and Time 120min
  Plasminogen (%)
Hb | Baseline, Time 15min, and Time 120min
  Hemoglobin (g/dl)
Platelets | Baseline, Time 15min, and Time 120min
  Platelets (G/l)
TP | Baseline, Time 15min, and Time 120min
  Prothrombin ratio (%)
aPTT ratio | Baseline, Time 15min, and Time 120min
  Activated Cephalin Time (sec)
Fibrinogen | Baseline, Time 15min, and Time 120min
  Fibrinogen (g/l)
Fibrin degradation products | Baseline, Time 15min, and Time 120min
  Fibrin degradation products (µg/l)
Plasmin-antiplasmin complex | Baseline, Time 15min, and Time 120min
  Plasmin-antiplasmin complex (µg/l)
Thrombin-antithrombin complex | Baseline, Time 15min, and Time 120min
  Thrombin-antithrombin complex (ng/ml)
Bleeding | Baseline, Time 15min, and Time 120min
  Bleeding (ml)
Transfusion of packs of red blood cells | Time 120min
  Number of packs of red blood cells
Transfusion of platelet concentrates | Time 120min
  Number of platelet concentrates
Transfusion of plasma | Time 120min
  volume of plasma (ml)
Transfusion of fibrinogen concentrate | Time 120min
  Amount (g) of fibrinogen concentrate

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No